CLINICAL TRIAL: NCT04904393
Title: Subanalysis in Patients With CARDIoLAMinopathy Enrolled to Retrospective and Observational Registy on Cardiac Contractility Modulation Therapy
Brief Title: Subanalysis in Patients With CARDIoLAMinopathy Enrolled to REPORT-CCM Registry
Acronym: CARDILAM-CCM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Monaldi Hospital (Other)
Responsible Party: Principal Investigator, Antonio D'Onofrio, Head of UOSD Elettrofisiologia Studio e Terapia delle Aritmie, Monaldi Hospital
Other Study IDs: CCM-002Mon
Record Dates: First submitted 2021-05-15; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Laminopathy; Lamin A/C Gene Mutation; Heart Failure
Keywords: Heart Failure; Cardiac Contyractility Modulation; Quality of Life
MeSH Terms: conditions — Laminopathies; Heart Failure | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Implant of the device for Cardiac Contractility Modulation (CCM) Therapy — The intervention is an implant of CCM therapy devices and it is similar to conventional dual chamber cardiac devices with only difference of to insert n 2 leads fixed in right ventricular septum

SUMMARY:
Observational, retrospective registry with acute and chronic endpoints

DETAILED DESCRIPTION:
This registry includes patients who have undergone CCM device implant and due to the presence of heart failure with reduced left ventricular systolic function and symptomatic despite optimal therapy, with LMNA-DCM etiology for to assess the impact on CCM therapy in term of improvemente of QoL and reduction HF hospitalizations

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female, aged 18 or older;
* chronic heart failure with symptomatic left ventricular systolic function (NYHA class II-IVa) with or without device already implanted (for example AICD, pace-maker);
* Appropriate and optimized medical therapy;
* Patient signed and dated informed consent form at enrollment;
* life expectancy> 1 year due to the absence of comorbidities that reduce the prognosis

Exclusion Criteria:

* absence of venous access available for implant;
* contraindication to the interventional procedure of CCM device implant (for example presence of Mechanical tricuspid vale);
* pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with standard indication to CCM therapy device implantation with Cardiolaminopahy aetiology and in HF status.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of QoL | 12 months
  Evaluation of the effect of CCM therapy on Quality of Life evaluated from the reduction of MLWHFQ score at FU post implant of CCM device compared to baseline.
Reduction of HF Hospitalizations and Emergency Ward accesses | 12 months
  Reduction of HF Hospitalizations and Emergency Ward accesses collected during the FU post implant of CCM device compared to number of Hospitalizations and Emergenncy Ward accesses collected 1 year before the implant of CCM therapy device
Improvement of Fuctional Capacity | 12 months
  Evaluation of the impact of CCM therapy on Functional Capacity evaluated from the gain of the distance travelled in the 6MWT at FU post implant of CCM therapy device compared to baseline

SECONDARY OUTCOMES:
Assess of HF biomarkers trends | 12 months
  Assess of HF biomarkers trends (laminine, NT-ProBNP, copeptine) during the FU compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Antonio D'Onofrio, MD, Study Director — Ao dei Colli - Monaldi Hospital
Locations (1):
- AO dei Colli - Monaldi Hospital, Naples, Italy